CLINICAL TRIAL: NCT04605003
Title: Effectiveness of Nasal Endoscope Sterilization Using a Novel Rig-S™ Device: A Randomized Controlled Trial
Brief Title: Effectiveness of Nasal Endoscope Sterilization Using a Novel Rig-S™ Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Azlina Ab Rani, Principal investigator, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Novel rig-S
Record Dates: First submitted 2020-10-16; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Sterility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The swabbing of the endoscopes are performed by a research assistant, and the end result is evaluated by the primary investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Autoclave (Active Comparator): The conventional autoclave is the gold standard of sterilising all medical equipments.
  Interventions: Device: Novel rig-S; Device: Conventional Autoclave machine
- Novel rig-S (Active Comparator): A novel devise used with the high level disinfectant
  Interventions: Device: Novel rig-S; Device: Conventional Autoclave machine

INTERVENTIONS:
Device: Novel rig-S — A new device created to hold the high level disinfectant and automatically indicate when sterilisation process has been completed
Device: Conventional Autoclave machine — The gold standard device to clean all medical instruments

SUMMARY:
This study compares the sterility of rigid nasoendoscopies after being sterilized with a conventional autoclave machine and a novel rig-S device that uses standard high level disinfectant

DETAILED DESCRIPTION:
There is a standard operating procedure in rigid endoscopy cleaning, and it is performed after each clinical examination. The conventional autoclave is no longer used in the setting of an otorhinolaryngology (ORL) clinic as it is cumbersome and takes a lot of time, and also only cleans one endoscope at a time. There is no standardisation or device that has been reported, and cross contamination has been reported previously. The overturn of patients in the ORL clinic is high, and most practitioners chooses high level disinfectant as a method of sterilising the endoscopes. However, there is no proper device to place these disinfectants in, and results in many cases of broken scopes and cross contamination.

This study compares the sterility of the rigid endoscopes after being sterilised by the high level disinfectant that is placed in a novel rig-S device with the gold standard conventional autoclave.

The investigators selected all the rigid endoscopes performed in our ORL clinic and randomised them before subjecting them for a swab test for bacterial and fungal, and also used a test kit to test the presence of Hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

All rigid endoscopes performed in ORL clinic

Exclusion Criteria:

Flexible endoscopes performed in ORL clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Microbial and Hepatitis B test | 3 days
  Rigid endoscopes are swabbed and tested using a hep-B kit

SECONDARY OUTCOMES:
Acidity level | 4 hours
  Acidity level of the high level disinfectant is tested for every 10 cycles of scope

CONTACTS AND LOCATIONS:
Overall Officials: Salina Husain, MMED, Study Director — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- Universiti Kebangsaan Malaysia, Cheras, Kuala Lumpur, Malaysia